CLINICAL TRIAL: NCT06353009
Title: Effect of a Single Ultra-Processed Meal on Myocardial Endothelial Function Assessed With Positron Emission Tomography
Acronym: SUPPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matthieu Pelletier-Galarneau, MD MSc (Other)
Responsible Party: Sponsor-Investigator, Matthieu Pelletier-Galarneau, MD MSc, Chief, division of nuclear medicine at Institut de cardiologie de Montreal, Montreal Heart Institute
Organization: Montreal Heart Institute (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: ICM 2021-2720
Record Dates: First submitted 2024-03-15; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Myocardial Endothelial Function

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: NOVA4 meal — NOVA (a name, not an acronym) is a food classification system divided into four groups, based on the level of processing.
  Group 4 - Ultra-processed foods. They are the ones that use many ingredients including food additives that improve palatability, processed raw materials (hydrogenated fats, modified starches, etc.) and ingredients that are rarely used in home cooking such as soy protein or mechanically separated meat. These foods are mainly of industrial origin and are characterized by a good pleasantness and the fact that they can be stored for a long time.
Other: NOVA1-3 meal — NOVA (a name, not an acronym) is a food classification system divided into four groups, based on the level of processing.
  Group 1 - Unprocessed or minimally processed foods (fruit, vegetables, eggs, meat, milk, etc.)
  Group 2 - Foods processed in the kitchen with the aim of extending their shelf life. In practice, these are ingredients to be used in the kitchen such as fats, aromatic herbs, etc. to be kept in jars or in the refrigerator to be able to use them later.
  Group 3 - Processed foods. These are the foods obtained by combining foods of groups 1 and 2 to obtain the many food products for domestic use (bread, jams, etc.) made up of a few ingredients

SUMMARY:
The objective of this study is to evaluate the effect of an ultra-processed meal on myocardial endothelial function using positron emission tomography (PET).

The proposed study is an open-label, randomized crossover clinical trial. Participants will be divided into 2 groups: half of the participants will consume a Mediterranean meal during the first experimental visit and an ultra-processed meal during the second, and vice versa for the other half. The order in which the meals will be consumed will be determined randomly.

This project will contribute to clarify the role of diet in the development and progression of coronary artery disease. The results obtained from this study may potentially demonstrate the harmful effect of ultra-processed foods, even in the short term, on coronary arteries.

DETAILED DESCRIPTION:
The proposed study is an open-label, randomized crossover trial. This design will allow participants to serve as their own controls. This is critical as there is some variability in response to vasodilators in the population, and by using this research design, we increase our ability to detect small changes. The study consists of 3 visits: a preliminary visit and two imaging visits. During the preliminary visit, the study will be explained to participants, and consent will be obtained. During the imaging visits, participants will consume a meal, and PET imaging will be completed 4 hours later. Half of the participants will consume the Mediterranean meal during the first visit and the ultra-processed meal during the second visit, and vice versa for the other participants. Randomization will determine the order in which the meals are consumed.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged between 18 and 50 years.
2. Absence of cardiovascular symptoms.
3. Ability to provide free and informed consent.

Exclusion Criteria:

1. Presence of cardiovascular disease.
2. Active smoking or within the past 12 months.
3. Hypertension (BP > 140/90 mmHg).
4. Renal failure (Creatinine clearance < 90 mL/min).
5. Type I or II diabetes.
6. Dyslipidemia (LDL ≥ 3.5 mmol/L or total cholesterol/HDL ratio ≥ 5.0).
7. Heart failure (Left ventricular ejection fraction < 50%).
8. Congenital heart disease.
9. Obesity (BMI > 35 kg/m2).
10. Uncontrolled asthma or chronic obstructive pulmonary disease (COPD).
11. History of severe allergy or reaction to adenosine or dipyridamole.
12. Second-degree type II or third-degree atrioventricular block.
13. Bradycardia with resting heart rate < 40 bpm.
14. Chronic alcoholism.
15. Substance abuse.
16. Claustrophobia.
17. Vegetarianism.
18. Use of statins or beta-blockers.
19. Food allergy preventing consumption of study meals.
20. Participation in this project would result in cumulative research study radiation dose > 50 mSv in the past 12 months.
21. Neurocognitive disorders or medication use affecting cognition.
22. Any condition that, in the opinion of the investigators, could compromise the subject's participation in the study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women excluded to avoir hormonal cycle variation in endothelial function.
Enrollment: 15 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Myocardial blood flow values (ml/min/g) at maximum dose of adenosine. | 4 hours after meal consumption
  The difference in maximum dose adenosine myocardial blood flow measured after consumption of ultra-processed (NOVA 4) and Mediterranean meals (NOVA 1-3) in healthy subjects.

SECONDARY OUTCOMES:
Myocardial blood flow values (ml/min/g) at rest and myocardial reserve. | 4 hours after meal consumption
  The difference in myocardial blood flow at rest and myocardial reserve, measured after ultra-processed (NOVA 4) and Mediterranean (NOVA1-3) meals in healthy subjects.
Myocardial blood flow values (ml/min/g) at intermediate dose of adenosine. | 4 hours after meal consumption
  The difference in myocardial blood flow at intermediate dose of adenosine, measured after ultra-processed (NOVA 4) and Mediterranean (NOVA 1-3) meals in healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Pelletier-Galarneau, Principal Investigator — Montreal Heart Institute
Locations (1):
- Matthieu Pelletier-Galarneau, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lucinian YA, Gagnon C, Latour E, Hamel V, Iglesies-Grau J, Nigam A, Harel F, Nozza A, Juneau M, Moubarac JC, Bherer L, Pelletier-Galarneau M. Effect of a single ultra processed meal on myocardial endothelial function, adenosine mediated effects and cognitive performances. Sci Rep. 2025 Aug 6;15(1):28671. doi: 10.1038/s41598-025-11734-z. PMID 40764338